CLINICAL TRIAL: NCT02657213
Title: Study of Minimed 640G Insulin Pump With SmartGuard in Prevention of Low Glucose Events in Adults With Type 1 Diabetes at Risk of Severe Hypoglycemia
Brief Title: Study of Insulin Pump in Prevention of Low Glucose Events in Adults With Type 1 Diabetes at Risk of Severe Hypoglycemia
Acronym: ALPPHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 38RC15.110
Record Dates: First submitted 2016-01-06; First posted 2016-01-15 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Diabetes, Type 1
Keywords: Diabetes, Type 1; Hypoglycemia; Insulin Infusion Systems
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimed 640G with smartguard activated (Experimental): Group "SmartGuard On": Patients will be equipped with a sensor augmented pump (SAP) therapy Minimed 640G insulin pump with SmartGuard activation
  Interventions: Device: Minimed 640G with smartguard activated
- Minimed 640G with smartguard off (Active Comparator): Group "SmartGuard Off" Patients will be equipped with a sensor augmented pump (SAP) therapy Minimed 640 insulin pump without SmartGuard activation
  Interventions: Device: Minimed 640G with smartguard off

INTERVENTIONS:
Device: Minimed 640G with smartguard activated — Patients will be equipped with a Minimed 640G insulin pump coupled with Enlite sensor with SmartGuard activation
  Other Names: Minimed 640G insulin Pump with Smartguard activation
  Arms: Minimed 640G with smartguard activated
Device: Minimed 640G with smartguard off — Patients will be equipped with Minimed 640G insulin pump coupled with Enlite glucose sensor without SmartGuard activation
  Other Names: Minimed 640G insulin Pump without activated Smartguard
  Arms: Minimed 640G with smartguard off

SUMMARY:
The main objective is to evaluate the efficacy of sensor augmented pump (SAP) therapy with MiniMed 640G with SmartGuard activation in preventing hypoglycemia events in comparison sensor augmented pump (SAP) therapy with Minimed 640G without SmartGuard activation in type 1 diabetic adults with an increased risk of hypoglycemia.

The study should show:

* A reduction in the number of severe hypoglycemia, fewer hypoglycemic events and a reduction in the time spent in hypoglycemia six months in any group compared to Baseline.
* A complete prevention of severe and not severe hypoglycemia in the pump group Minimed 640G + Enlite sensor with SmartGuard activation

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or insulin-dependent diabetic patients
* Patients treated with subcutaneous insulin pump with at least 2 episodes of severe hypoglycemia within 12 months before the study enrollment
* Affiliation to the french social security system or equivalent
* People who signed the consent form

Exclusion Criteria:

* Patient who have difficulty to understand the French language
* Patient can not be raised to the use of an insulin pump, or a glucose sensor
* Patient visually impaired
* Patient hard of hearing
* Pregnant woman or woman having a project of pregnancy within 6 months
* Persons referred to in Articles L1121-5 to L1121-8 CSP: pregnant woman, woman in labor, breastfeeding women, persons deprived of their liberty by judicial or administrative decision, person under a legal protection measure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the Minimed 640G insulin pump with Smartguard activation in preventing the number of severe and non-severe hypoglycaemia in patients with diabetes type 1 at risk of severe hypoglycemia | 6 months
  Number of events of hypoglycemia (severe and non-severe)

SECONDARY OUTCOMES:
Assessment of Improving of overall glycemic control with SmartGuard activation in type 1 diabetic patients at risk of severe hypoglycemia | 6 months
  Comprehensive metabolic evaluation data and evaluation data of severe hypoglycaemic risk
Assessment of the quality of life of patients with smartguard activation | 6 months
  Quality of Life Questionnaire
Assessment of the number of adverse events | 6 months
  Assessment of the safety of the sensor augmented pump therapy with the Mimimed 640G insulin pump coupled with a 640G Minimed Enlite sensor with Smart Guard as compare to sensor augmented pump therapy with the Mimimed 640G insulin pump coupled with a 640G Minimed Enlite sensor without Smart Guard activation (Decompensated ketoacidosis, Hospitalization related to severe hypoglycemia or frequent hypoglycemia or moderate decompensation, Materiovigilance data, Collection and monitoring of serious adverse events and non-serious)
Study of average cost per patient for each therapeutic strategy supported from the point of view of society | 6 months
  An average cost per patient will be calculated for each strategy. The horizon time is 6 months from randomization of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine LABLANCHE, MD, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - Grenoble University Hospital, Grenoble
  - Montpellier University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergenstal RM, Klonoff DC, Garg SK, Bode BW, Meredith M, Slover RH, Ahmann AJ, Welsh JB, Lee SW, Kaufman FR; ASPIRE In-Home Study Group. Threshold-based insulin-pump interruption for reduction of hypoglycemia. N Engl J Med. 2013 Jul 18;369(3):224-32. doi: 10.1056/NEJMoa1303576. Epub 2013 Jun 22. PMID 23789889
- [Background] European User Evaluation of the MiniMed® 640G system. Poster session at the American Diabetes Association (ADA) 75th Scientific Sessions on Sunday, June 7 2015. Boston Convention and Exhibition Center.